CLINICAL TRIAL: NCT04029688
Title: A Phase I/II, Multicenter, Open-Label, Multi-Arm Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Activity of Idasanutlin in Combination With Either Chemotherapy or Venetoclax in the Treatment of Pediatric and Young Adult Patients With Relapsed/Refractory Acute Leukemias or Solid Tumors
Brief Title: A Study Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Activity of Idasanutlin in Combination With Either Chemotherapy or Venetoclax in Treatment of Pediatric and Young Adult Participants With Relapsed/Refractory Acute Leukemias or Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated by the sponsor based on insufficient tolerability and efficacy to proceed beyond Part 1b.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO40871; 2018-004579-11 (EudraCT Number)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Neuroblastoma; Solid Tumors
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neuroblastoma | interventions — RG7388; venetoclax; Cyclophosphamide; Topotecan; fludarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation: Solid Tumors: Idasanutlin Single Agent (Experimental)
  Interventions: Drug: Idasanutlin
- Neuroblastoma: Idasanutlin + Venetoclax (Experimental)
  Interventions: Drug: Idasanutlin; Drug: Venetoclax
- Neuroblastoma: Idasanutlin + Cyclophosphamide + Topotecan (Experimental)
  Interventions: Drug: Idasanutlin; Drug: Cyclophosphamide; Drug: Topotecan
- AML: Idasanutlin + Venetoclax (Experimental)
  Interventions: Drug: Idasanutlin; Drug: Venetoclax; Drug: Intrathecal Chemotherapy
- AML: Idasanutlin + Fludarabine + Cytarabine (Experimental)
  Interventions: Drug: Idasanutlin; Drug: Fludarabine; Drug: Cytarabine; Drug: Intrathecal Chemotherapy
- ALL: Idasanutlin + Venetoclax (Experimental)
  Interventions: Drug: Idasanutlin; Drug: Venetoclax; Drug: Intrathecal Chemotherapy

INTERVENTIONS:
Drug: Idasanutlin — Idasanutlin will be administered as an oral medication once daily on Days 1-5 of a 28-day cycle.
  Other Names: RG7388
Drug: Venetoclax — Venetoclax will be administered orally at the adult dose equivalent (adjusted by body weight) of 400 milligrams (mg) in participants with neuroblastoma and the adult dose equivalent of 600 mg in participants with leukemia.
  Other Names: RG7601; GDC-0199; ABT-199
  Arms: ALL: Idasanutlin + Venetoclax; AML: Idasanutlin + Venetoclax; Neuroblastoma: Idasanutlin + Venetoclax
Drug: Cyclophosphamide — Cyclophosphamide will be administered once daily on Days 1-5 of each 28-day cycle at 250 milligrams per meter squared of body surface area (mg/m^2) as an intravenous (IV) infusion.
  Arms: Neuroblastoma: Idasanutlin + Cyclophosphamide + Topotecan
Drug: Topotecan — Topotecan will be administered once daily on Days 1-5 of each 28-day cycle at 0.75 mg/m^2 as an IV infusion.
  Arms: Neuroblastoma: Idasanutlin + Cyclophosphamide + Topotecan
Drug: Fludarabine — Fludarabine will be administered once daily on Days 1-5 of each 28-day treatment cycle at 30 mg/m^2 as an IV infusion.
  Arms: AML: Idasanutlin + Fludarabine + Cytarabine
Drug: Cytarabine — Cytarabine will be administered once daily on Days 1-5 of each 28-day treatment cycle at 2000 mg/m^2 as an IV infusion.
  Arms: AML: Idasanutlin + Fludarabine + Cytarabine
Drug: Intrathecal Chemotherapy — All participants with leukemia, irrespective of arm, will receive intrathecal chemotherapy on Day 1 of each 28-day treatment cycle. Intrathecal chemotherapy will consist of either single-agent cytarabine or methotrexate, or a combination of methotrexate, cytarabine, and hydrocortisone, at appropriate age-based dosing as specified in the protocol.
  Arms: ALL: Idasanutlin + Venetoclax; AML: Idasanutlin + Fludarabine + Cytarabine; AML: Idasanutlin + Venetoclax

SUMMARY:
This is a Phase I/II, multicenter, open-label, multi-arm study designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of idasanutlin, administered as a single agent or in combination with chemotherapy or venetoclax, in pediatric and young adult participants with acute leukemias or solid tumors.

This study is divided into three parts: Part 1 will begin with dose escalation of idasanutlin as a single agent in pediatric participants with relapsed or refractory solid tumors to identify the maximum tolerated dose (MTD)/maximum administered dose (MAD) and to characterize dose-limiting toxicities (DLTs). Following MTD/MAD identification, three separate safety run-in cohorts in neuroblastoma, acute myeloid leukemia (AML), and acute lymphoblastic leukemia (ALL) will be conducted to identify the recommended Phase 2 dose (RP2D) of idasanutlin in each combination, with chemotherapy or venetoclax. Part 2 will evaluate the safety and early efficacy of idasanutlin in combination with chemotherapy or venetoclax in newly enrolled pediatric and young adult participants in neuroblastoma, AML,and ALL cohorts at idasanutlin RP2D. Part 3 will potentially be conducted as an additional expansion phase of the idasanutlin combination cohorts in neuroblastoma, AML, or ALL for further response and safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* The participants ages are < 18 for part 1a, < 30 for Parts 1b. 2 and 3
* Study Part 1 (single-agent therapy dose escalation): histologically confirmed diagnosis of neuroblastoma or other solid tumor that has progressed or recurred despite standard therapy, and for which there is no therapy proven to prolong survival with an acceptable quality of life
* Study Part 1 (combination safety run-in), Study Part 2 (initial expansion), and Study Part 3 (additional expansion): histologically confirmed diagnosis of neuroblastoma, AML, or precursor-B ALL that has progressed or recurred despite, or is refractory to, standard therapy
* Adequate performance status: Participants <16 years of age: Lansky greater than or equal to (≥)50%; Patients ≥16 years of age: Karnofsky ≥50%
* Adequate end-organ function, as defined in the protocol
* For females of childbearing potential: agreement to remain abstinent, use contraception, agreement to refrain from donating eggs. Females must remain abstinent or use two methods of contraception with a failure rate of <1% per year during the treatment and follow-up period (variable depending on the combination agent) or in accordance with national prescribing information guidance regarding abstinence, contraception
* For males: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm, with a female partner of childbearing potential or pregnant female partner, males must remain abstinent or use a condom during the treatment period and for follow-up period (variable, depending on the combination agent) or in accordance with national prescribing information guidance regarding abstinence, contraception

Additional Inclusion Criteria for Participants with Solid Tumors (including Neuroblastoma)

* At least one evaluable or measurable radiological site of disease as defined by standard criteria for the participant's tumor type, or measurable bone marrow disease by morphology
* Adequate hematologic end-organ function, as defined in the protocol
* Tumor tissue from relapsed disease

Additional Inclusion Criteria for Patients with Leukemia

* Bone marrow with ≥5% lymphoblasts by morphologic assessment at screening
* Available bone marrow aspirate or biopsy from screening

Exclusion Criteria:

* Primary Central Nervous System (CNS) tumors
* Symptomatic CNS metastases that result in a neurologically unstable clinical state or require increasing doses of corticosteroids or local CNS-directed therapy to control the CNS disease
* CNS3 leukemia
* Acute promyelocytic leukemia
* White blood cell count >50 × 10^9 cells/Liter (L)
* Down syndrome, Li-Fraumeni syndrome, history of severe aplastic anemia, or any known bone marrow failure predisposition syndrome
* Burkitt-type acute lymphoblastic leukemia
* T-cell lymphoblastic leukemia
* Prior treatment with a MDM2 antagonist
* Prior treatment with venetoclax (if potential for enrollment in a venetoclax arm)
* Infection considered by the investigator to be clinically uncontrolled or of unacceptable risk to the participant
* Any uncontrolled medical condition or other identified abnormality that precludes the patient's safe participation in and completion of the study
* Systemic anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to initiation of study treatment
* Treatment with monoclonal antibodies, antibody drug conjugates, or cellular therapy for anti-neoplastic intent within 30 days prior to initiation of study treatment
* I-131 meta-iodobenzylguanidine (MIBG) therapy within 6 weeks prior to initiation of study treatment
* Myeloablative therapy with autologous or allogeneic hematopoietic stem cell rescue within 100 days of study treatment initiation
* Immunosuppressive therapy for treatment of graft-versus-host disease within 2 weeks of study treatment initiation
* Radiotherapy within 3 weeks prior to study treatment initiation
* Specific restrictions are applicable for patients treated with drugs interacting with CYP2C8, CYP3A4, OATP1B1/B3, and P-gp
* Received anti-coagulant or anti-platelet agent within 7 days or 5 half-lives prior to study treatment initiation
* Underwent major surgical procedure within 21 days of study treatment initiation, or anticipate need for major surgical procedure during the course of the study

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (5):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Lucile Packard Children's Hospital at Stanford University; Thoracic Oncology, Palo Alto, California
  - Arnold Palmer Hosp-Children, Orlando, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Alberta Children'S Hospital, Calgary, Alberta, Canada
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
- Prinses Maxima Centrum, Utrecht, Netherlands
- Spain (2):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - The Royal Victoria Infirmary; Paediatric and Adolescent Oncology Unit, Newcastle upon Tyne
  - Royal Marsden Hospital; Pediatric Unit, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Rubio-San-Simon A, Marshall LV, Doz F, Mora J, Bielamowicz K, Corradini N, Langevin AM, Narendran A, Smith AA, Zwaan CM, Gho D, Cardenas A, Fowler S, Guizani C, Breton V, Wulff B, Bernardi R, Trippett T, Campbell-Hewson Q. Idasanutlin in Combination with Chemotherapy or Venetoclax in Pediatric and Young Adult Patients with Relapsed/Refractory Solid Tumors (iMATRIX Idasa): Results of a Phase I/II, Multicenter, Multi-arm Study. Target Oncol. 2025 Dec 11. doi: 10.1007/s11523-025-01186-w. Online ahead of print. PMID 41379293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with relapsed/refractory solid tumors took part in the study across 12 investigative sites in 6 countries (United States, Spain, United Kingdom, France, Canada, and Netherlands) from January 27, 2020 to May 6, 2024.
Pre-assignment Details: Study was divided into 3 parts. Part 1a: Single agent idasanutlin dose escalation in pediatric participants with solid tumors. Part 1b: Combination safety run-in in participants with neuroblastoma/acute leukemia. Part 2: Early efficacy in participants with neuroblastoma/acute leukemia. Part 3: Expansion cohorts in participants with neuroblastoma/acute leukemia. Leukemia cohorts in Part 1b & all cohorts in Part 2 & Part 3 were never initiated due to early termination of the study by the sponsor.
Groups:
- Part 1a: Idasanutlin 2 Milligrams/Kilograms (mg/kg): Participants with solid tumors received idasanutlin 2 mg/kg orally once daily (QD) on Days 1-5 of each 28-day cycle until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1a: Idasanutlin 3 mg/kg: Participants with solid tumors received idasanutlin 3 mg/kg orally QD on Days 1-5 of each 28-day cycle until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1a: Idasanutlin 4.5 mg/kg: Participants with solid tumors received idasanutlin 4.5 mg/kg orally QD on Days 1-5 of each 28-day cycle until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1a: Idasanutlin 6.4 mg/kg: Participants with solid tumors received idasanutlin 6.4 mg/kg orally QD on Days 1-5 of each 28-day cycle until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1a: Idasanutlin 8 mg/kg: Participants with solid tumors received idasanutlin 8 mg/kg orally QD on Days 1-5 of each 28-day cycle until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1b: Idasanutlin (2.8 mg/kg) +Chemotherapy: Participants with neuroblastoma received idasanutlin 2.8 mg/kg orally in combination with cyclophosphamide 200 milligrams per square meter (mg/m^2) and topotecan 0.6 mg/m^2 as an IV infusion QD on Days 1-5 of each 28-day cycle. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1b: Idasanutlin (3.6 mg/kg) +Chemotherapy: Participants with neuroblastoma received idasanutlin, 3.6 mg/kg orally, in combination with cyclophosphamide 250 mg/m^2 and topotecan 0.75 mg/m^2 as an IV infusion QD on Days 1-5 of each 28-day cycle. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax: Participants with neuroblastoma (first 3) received idasanutlin, 3.6 mg/kg orally QD on Days 1-5, in combination with venetoclax 400 milligrams (mg) adult dose equivalent (adjusted by body weight) on Days 1-28 of each 28-day cycle. After the first three participants were treated, the schedule was modified as idasanutlin, 3.6 mg/kg orally QD on Days 1-5 and venetoclax 400 mg (adult dose equivalent) on Days 1-14 of a each 28-day cycle for the next 3 participants enrolled in this arm. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
Period: Overall Study
Arm/Group | Part 1a: Idasanutlin 2 Milligrams/Kilograms (mg/kg) | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg | Part 1b: Idasanutlin (2.8 mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6 mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Started | 8 | 3 | 6 | 3 | 6 | 3 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 3 | 6 | 3 | 6 | 3 | 3 | 6
Not completed — Death | 8 | 3 | 6 | 2 | 5 | 0 | 2 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all enrolled participants in the study, regardless of whether they were dosed.
Groups:
- Part 1a: Idasanutlin 2 mg/kg: Participants with solid tumors received idasanutlin 2 mg/kg QD on Days 1-5 of each 28-day cycle until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1b: Idasanutlin (2.8 mg/kg) +Chemotherapy: Participants with neuroblastoma received idasanutlin 2.8 mg/kg orally in combination with cyclophosphamide 200 mg/m^2 and topotecan 0.6 mg/m^2 as an IV infusion QD on Days 1-5 of each 28-day cycle. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax: Participants with neuroblastoma (first 3) received idasanutlin, 3.6 mg/kg orally QD on Days 1-5, in combination with venetoclax 400 mg adult dose equivalent (adjusted by body weight) on Days 1-28 of each 28-day cycle. After the first three participants were treated, the schedule was modified as idasanutlin, 3.6 mg/kg orally QD on Days 1-5 and venetoclax 400 mg (adult dose equivalent) on Days 1-14 of a each 28-day cycle for the next 3 participants enrolled in this arm. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg | Part 1b: Idasanutlin (2.8 mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6 mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax | Total
Number analyzed (Participants) | 8 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (5.0) | 11.3 (3.2) | 7.3 (3.9) | 15.0 (1.7) | 11.5 (5.0) | 15.0 (11.4) | 5.3 (1.2) | 8.0 (3.8) | 9.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 2 | 1 | 3 | 1 | 1 | 2 | 16
  Male | 3 | 2 | 4 | 2 | 3 | 2 | 2 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 6
  Not Hispanic or Latino | 3 | 1 | 2 | 3 | 4 | 3 | 2 | 2 | 20
  Unknown or Not Reported | 3 | 1 | 3 | 0 | 2 | 0 | 0 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
  White | 4 | 2 | 2 | 3 | 3 | 3 | 1 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 3 | 0 | 3 | 0 | 1 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Part 1a and 1b: Number of Participants With Adverse Events (AEs) and Severity of AEs Determined According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5 (NCI CTCAE v5.0)
Description: An AE is any untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. AEs were graded as per NCI CTCAE v5.0. Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living; Grade 4=Life-threatening consequences/urgent intervention indicated; Grade 5=Death related to adverse event.
Time Frame: From screening up to 30 days after study treatment discontinuation (approximately 7 months)
Population: Safety evaluable (SE) population included all participants who received any amount of the study treatment, whether prematurely withdrawn from the study or not.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy: Participants with neuroblastoma received idasanutlin 2.8 mg/kg orally in combination with cyclophosphamide 200 mg/m^2 and topotecan 0.6 mg/m^2 as an IV infusion QD on Days 1-5 of each 28-day cycle. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
- Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy: Participants with neuroblastoma received idasanutlin, 3.6 mg/kg orally, in combination with cyclophosphamide 250 mg/m^2 and topotecan 0.75 mg/m^2 as an IV infusion QD on Days 1-5 of each 28-day cycle. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 8 | 3 | 6 | 3 | 6 | 3 | 3 | 6
Participants
  AEs, Any Grade | 8 | 3 | 6 | 3 | 6 | 3 | 3 | 6
  AEs, Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AEs, Grade 3 | 2 | 1 | 3 | 2 | 1 | 0 | 0 | 3
  AEs, Grade 4 | 5 | 2 | 3 | 1 | 5 | 3 | 3 | 1
  AEs, Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Parts 1a and 1b: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLTs were assessed for single-agent idasanutlin and idasanutlin in combination with chemotherapy or venetoclax. A DLT was defined as any AE that occurred during the DLT assessment window and was assessed by the investigator as related or possibly related to idasanutlin. An AE is an untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. Following events were considered to be DLTs: any treatment-related death; elevation of serum hepatic transaminase; severe liver injury, in the absence of cholestasis or other causes of hyperbilirubinemia; any non-hematologic toxicity Grade ≥3; nausea, vomiting, and/or diarrhea if Grade 3 severity lasts > than 24 hours after initiation of supportive care measures or if Grade 4 or higher; hematologic toxicity; any related event that results in a dose delay beyond Day 42.
Time Frame: Cycle 1 (one cycle is 28 days)
Population: DLT-evaluable population included all participants enrolled in Part 1 who either completed at least 80% of the prescribed dose of idasanutlin and the DLT observation window in Cycle 1 OR have experienced a DLT in Cycle 1 of the dose-escalation phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 8 | 3 | 6 | 3 | 6 | 3 | 3 | 6
Participants | 0 | 0 | 1 | 0 | 4 | 1 | 2 | 0

3. Primary Outcome: Part 1b: Objective Response Rate (ORR) in Participants With TP53 Wild-Type (WT) Neuroblastoma Assessed According to International Neuroblastoma Response Criteria (INRC)
Description: ORR was defined as the percentage of participants with complete response (CR) or partial response (PR) at any time during study treatment, on 2 consecutive occasions ≥ 4 weeks apart, as determined by the investigator per INRC. Primary tumor: CR = <10 millimeters (mm) residual soft tissue at primary site and complete resolution of meta-iodobenzylguanidine (MIBG) or fluorodeoxyglucose-positron emission tomography (FDG-PET) uptake at primary site. PR = ≥ 30% decrease in longest diameter of primary site and MIBG or FDG-PET uptake at primary site stable, improved, or resolved. Soft tissue & bone metastases: CR = resolution of all disease sites; PR = ≥30% decrease in sum of non-primary target lesions, with no new lesions or ≥50% reduction in MIBG score or in number of FDG-PET-avid bone lesions; Bone marrow: CR = no tumor infiltration on reassessment.
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: Participants in the SE population who had TP53 WT tumor as assessed by central testing were analyzed for this outcome measure. SE Population included all participants who received any amount of the study treatment, whether prematurely withdrawn from the study or not. Percentages have been rounded off to the nearest decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 2 | 3 | 4
percentage of participants | 0 [0.0 to 84.19] | 33.3 [0.84 to 90.57] | 0 [0.0 to 60.24]

4. Primary Outcome: Parts 2 and 3: ORR in Participants With TP53 WT Neuroblastoma Assessed According to INRC
Description: ORR was defined as the percentage of participants with CR or PR at any time during study treatment, on 2 consecutive occasions ≥ 4 weeks apart, as determined by the investigator per INRC. Primary tumor: CR = <10 mm residual soft tissue at primary site and complete resolution of MIBG or FDG-PET uptake at primary site. PR = ≥ 30% decrease in longest diameter of primary site and MIBG or FDG-PET uptake at primary site stable, improved, or resolved. Soft tissue & bone metastases: CR = resolution of all disease sites; PR = ≥30% decrease in sum of non-primary target lesions, with no new lesions or ≥50% reduction in MIBG score or in number of FDG-PET-avid bone lesions; Bone marrow: CR = no tumor infiltration on reassessment.
Time Frame: Up to approximately 29 months
Population: The study was terminated before initiation of Parts 2 and 3 as per sponsor's decision. Hence no data were collected, and this outcome measure was not assessed or analyzed.
Groups:
- Part 2 (Neuroblastoma): Participants with neuroblastoma were planned to be enrolled in various cohorts in Part 2. Participants with neuroblastoma were to receive idasanutlin in combination with cyclophosphamide 250 mg/m^2 and topotecan 0.75 mg/m^2 on Days 1-5 of each 28-day cycle or venetoclax 400 mg.
- Part 3: Expansion (Neuroblastoma): Potential expansion of idasanutlin combination cohorts for participants with TP53 WT neuroblastoma from Parts 1b and 2 meeting the pre-defined efficacy criteria were planned to be initiated in Part 3.
Arm/Group | Part 2 (Neuroblastoma) | Part 3: Expansion (Neuroblastoma)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Parts 2 and 3: Complete Remission Rate (CRR) in Participants With TP53 WT Leukemia
Description: CRR was defined as the percentage of participants with morphologic complete remission (CR), complete remission with incomplete blood count recovery (CRi), or complete remission with incomplete platelet count recovery (CRp) within 2 cycles of study treatment. CR=Bone marrow blasts <5% (AML) and no evidence of circulating blasts, must be <1% (ALL); absence of blasts with Auer rods (AML); absence of extramedullary disease; absolute neutrophil count (ANC) >1.0*10^9/liter (L) [1000/microliter (µL)]; platelet count > 100*10^9/L (100,000/µL); independence of transfusions for a minimum of 1 week (AML and ALL). CRi= All CR criteria except for ANC <1.0*10^9/L[1000/µL] or insufficient recovery of platelet count <100* 10^9/L [100,000/µL] (AML and ALL). CRp=All CR criteria except for ANC >1.0*10^9/L[1000/µL]) or but with insufficient recovery of platelet (<100* 10^9/L [100,000/µL]) (ALL).
Time Frame: Up to Cycle 2 (cycle length=28 days) (approximately 8 weeks)
Population: as for outcome 4
Groups:
- Part 2 (Leukemia): Participants with acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) were planned to be enrolled in various cohorts in Part 2. Participants with AML were to receive idasanutlin plus fludarabine 30 mg/m^2 and high dose cytarabine 2000 mg/m^2 (FLA) on Days 1-5 of each 28-day cycle. Participants with ALL were to receive idasanutlin plus venetoclax 600 mg on Days 1-5 of each 28-day cycle.
- Part 3: Expansion (Leukemia): Potential expansion of idasanutlin combination cohorts for participants with TP35 WT AML or ALL from Parts 1b and 2 meeting the pre-defined efficacy criteria were planned to be initiated in Part 3.
Arm/Group | Part 2 (Leukemia) | Part 3: Expansion (Leukemia)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Parts 2 and 3: Minimal Residual Disease (MRD) - Negative Rate in Participants With ALL
Description: MRD - negative rate was defined as percentage of participants with ALL who have an MRD value < 0.01%, as measured by next-generation sequencing (NGS), within 2 cycles of study treatment.
Time Frame: Up to Cycle 2 (cycle length=28 days) (approximately 8 weeks)
Population: as for outcome 4
Groups:
- Part 2 (ALL): Participants with ALL were planned to be enrolled in Part 2 to receive idasanutlin plus venetoclax 600 mg on Days 1-5 of each 28-day cycle.
- Part 3: Expansion (ALL): Potential expansion of idasanutlin combination cohorts for participants with TP35 WT ALL from Parts 1b and 2 meeting the pre-defined efficacy criteria were planned to be initiated in Part 3.
Arm/Group | Part 2 (ALL) | Part 3: Expansion (ALL)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Part 1a: Clinical Benefit Rate (CBR) in Participants With Solid Tumors From SE Population Assessed According to Response Evaluation Criteria Version 1.1 (RECIST v1.1) or INRC
Description: CBR was defined as the percentage of participants achieving confirmed CR, PR, or stable disease (SD) on 2 consecutive occasions ≥4 weeks apart during the total study period. Per RECIST, CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference smallest sum on study. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference smallest sum on study (nadir), including baseline. Participants who had neuroblastoma were assessed by INRC. CR and PR per INRC were defined as outlined in the description for Part 1b: ORR outcome measure (OM).
Time Frame: From screening (maximum 28 days) up to Cycle 5 (cycle length=28 days)
Population: SE population included all participants who received any amount of the study treatment, whether prematurely withdrawn from the study or not. Percentages have been rounded off to the nearest decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg
Number analyzed (Participants) | 8 | 3 | 6 | 3 | 6
percentage of participants | 12.5 [0.32 to 52.65] | 33.3 [0.84 to 90.57] | 0 [0.0 to 45.93] | 66.7 [9.43 to 99.16] | 0 [0.0 to 45.93]

8. Secondary Outcome: Part 1b: CBR in Participants With Neuroblastoma From SE Population Assessed According to INRC
Description: CBR=percentage of participants with CR, PR, or SD on 2 consecutive occasions ≥ 4 weeks apart per INRC. Primary tumor: CR=residual soft tissue at primary site is <10 mm, with complete resolution of MIBG/FDG-PET uptake; PR= ≥30% decrease in longest diameter (LD) of primary site, with stable/improved MIBG/FDG-PET uptake; SD=Insufficient shrinkage for PR/increase for PD. PD= >20% increase in LD from smallest sum & minimum 5 mm increase in LD. Soft tissue & bone metastases: CR=resolution of all disease sites; PR= ≥30% decrease in sum of non-primary target lesions, with no new lesions or ≥50% reduction in MIBG score or in number of FDG-PET-avid bone lesions; PD=new soft tissue lesions per CT/MRI or MIBG/FDG-PET avid bone site; SD=no sufficient change in non-primary lesions. Bone marrow: CR=no tumor infiltration on reassessment; PD=new tumor infiltration >5% or infiltration increased >2-fold with >20% tumor infiltration; SD=persistent infiltration at >5% without meeting other criteria.
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 33.3 [0.84 to 90.57] | 33.3 [0.84 to 90.57] | 0 [0.0 to 45.93]

9. Secondary Outcome: Part 1b: CBR in Participants With TP53 WT Neuroblastoma Assessed According to INRC
Description: CBR=percentage of participants with CR, PR, or SD on 2 consecutive occasions ≥ 4 weeks apart per INRC. Primary tumor: CR=residual soft tissue at primary site is <10 mm, with complete resolution of MIBG/FDG-PET uptake; PR= ≥30% decrease in longest diameter (LD) of primary site, with stable/improved MIBG/FDG-PET uptake; SD=Insufficient shrinkage for PR or increase for PD. PD= >20% increase in LD from smallest sum & minimum 5 mm increase in LD. Soft tissue & bone metastases: CR=resolution of all disease sites; PR= ≥30% decrease in sum of non-primary target lesions, with no new lesions or ≥50% reduction in MIBG score or in number of FDG-PET-avid bone lesions; PD=new soft tissue lesions per CT/MRI or MIBG/FDG-PET avid bone site; SD=no sufficient change in non-primary lesions. Bone marrow: CR=no tumor infiltration on reassessment; PD=new tumor infiltration >5% or infiltration increased >2-fold with >20% tumor infiltration; SD=persistent infiltration at >5% without meeting other criteria.
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 2 | 3 | 4
percentage of participants | 50.0 [1.26 to 98.74] | 33.3 [0.84 to 90.57] | 0 [0.0 to 60.24]

10. Secondary Outcome: Part 1a: Duration of Response (DOR) in Participants With Solid Tumors From SE Population Assessed According to RECIST v1.1 or INRC
Description: DOR was defined as the time from the first tumor assessment that supports a participant's objective response (CR or PR) to the time of PD or death from any cause (whichever occurs first), as determined by the investigator using RECIST v1.1 or INRC. Per PRECIST, CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference smallest sum on study (nadir), including baseline. Participants who had neuroblastoma were assessed by INRC. CR/PR/PD were defined per INRC as outlined in the description for the Part 1b: CBR OM.
Time Frame: From screening (maximum 28 days) up to Cycle 5 (cycle length=28 days)
Population: SE population included all participants who received any amount of the study treatment, whether prematurely withdrawn from the study or not. DOR was only evaluated in participants who achieved an objective response (CR or PR).
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 1b: DOR in Participants With Neuroblastoma From SE Population Assessed According to INRC
Description: DOR=time from the first tumor assessment that supports a participant's objective response (CR or PR) to the time of PD or death from any cause (whichever occurs first), as determined by the investigator using INRC for participants with neuroblastoma. Primary tumor: CR=residual soft tissue at primary site is <10 mm, with complete resolution of MIBG/FDG-PET uptake; PR= ≥30% decrease in LD of primary site and MIBG or FDG-PET uptake at primary site stable, improved, or resolved; PD= >20% increase in LD from smallest sum & minimum 5 mm increase in LD. Soft tissue & bone metastases: CR = resolution of all disease sites; PR = ≥30% decrease in sum of non-primary target lesions, with no new lesions or ≥50% reduction in MIBG score or in number of FDG-PET-avid bone lesions; PD=new soft tissue lesions per CT/MRI or MIBG/FDG-PET avid bone site. Bone marrow: CR=no tumor infiltration on reassessment; PD=new tumor infiltration >5% or infiltration increased >2-fold with >20% tumor infiltration.
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 0 | 1 | 0
months |  | 4.5 [NA to NA] — Since only one participant showed response upper and lower limit of 95% CI were not evaluable. |

12. Secondary Outcome: Part 1b: DOR in in Participants With TP53 WT Neuroblastoma Assessed According to INRC
Description: as for outcome 11
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: Participants in the SE population who had TP53 WT tumor as assessed by central testing were analyzed for this outcome measure. SE Population included all participants who received any amount of the study treatment, whether prematurely withdrawn from the study or not. DOR was only evaluated in participants who achieved an objective response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 0 | 1 | 0
months |  | 4.5 [NA to NA] — Since only one participant showed response upper and lower limit of 95% CI were not evaluable. |

13. Secondary Outcome: Part 1a: Progression Free Survival (PFS) in Participants With Solid Tumors From SE Population Assessed According to RECIST v1.1 or INRC
Description: PFS was defined as the time from initiation of study drug to the first documented occurrence of PD or death from any cause (whichever occurs first), as determined by the investigator using RECIST or INRC. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference smallest sum on study (nadir), including baseline. Participants who had neuroblastoma were assessed by INRC. PD per INRC: Primary tumor = >20% increase in LD from smallest sum & minimum 5 mm increase in LD; Soft tissue & bone metastases = new soft tissue lesions per CT/MRI or MIBG/FDG-PET avid bone site; Bone marrow = new tumor infiltration >5% or infiltration increased >2-fold with >20% tumor infiltration.
Time Frame: From screening (maximum 28 days) up to Cycle 5 (cycle length=28 days)
Population: SE population included all participants who received any amount of the study treatment, whether prematurely withdrawn from the study or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg
Number analyzed (Participants) | 8 | 3 | 6 | 3 | 6
months | 0.8 [0.7 to 1.3] | 0.9 [0.9 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 0.8 [0.8 to 0.9] | 3.5 [2.8 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 1.9 [0.8 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events.

14. Secondary Outcome: Part 1b: PFS in Participants With Neuroblastoma From SE Population Assessed According to INRC
Description: PFS was defined as the time from initiation of study drug to the first documented occurrence of PD or death from any cause (whichever occurs first), as determined by the investigator using INRC for participants with neuroblastoma. Primary tumor: PD= >20% increase in LD from smallest sum & minimum 5 mm increase in LD. Soft tissue & bone metastases: PD=new soft tissue lesions per CT/MRI or MIBG/FDG-PET avid bone site. Bone marrow: PD=new tumor infiltration >5% or infiltration increased >2-fold with >20% tumor infiltration.
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 3 | 3 | 6
months | 1.9 [1.8 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 1.8 [1.6 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 1.7 [1.0 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events.

15. Secondary Outcome: Part 1b: PFS in Participants With TP53 WT Neuroblastoma Assessed According to INRC
Description: as for outcome 14
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: Participants in the SE population who had TP53 WT tumor as assessed by central testing were analyzed for this outcome measure. SE Population included all participants who received any amount of the study treatment, whether prematurely withdrawn from the study or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 2 | 3 | 4
months | NA [1.8 to NA] — The Median & upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 1.8 [1.6 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 1.7 [1.5 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events.

16. Secondary Outcome: Parts 1a and 1b: Overall Survival (OS) in SE Population
Description: OS was defined as the time from initiation of the study drug to death from any cause. Estimates for median OS were computed using Kaplan-Meier methodology
Time Frame: Up to approximately 29 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 8 | 3 | 6 | 3 | 6 | 3 | 3 | 6
months | 5.6 [2.1 to 20.8] | 12.5 [1.1 to NA] — Because of the small sample size, there is not enough information to construct a reliable upper confidence limit of the 95% CI for median survival using the applied Kaplan-Meier methodology. | 3.6 [2.3 to 9.8] | 16.4 [7.2 to NA] — Because of the small sample size, there is not enough information to construct a reliable upper confidence limit of the 95% CI for median survival using the applied Kaplan-Meier methodology. | 5.4 [3.4 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | NA [NA to NA] — The median and upper and lower limit of the 95% CI was not estimable because there was an insufficient number of events. | 3.2 [1.6 to NA] — Because of the small sample size, there is not enough information to construct a reliable upper confidence limit of the 95% CI for median survival using the applied Kaplan-Meier methodology. | NA [2.9 to NA] — Because of the small sample size, there is not enough information to construct a reliable upper confidence limit of the 95% CI for median survival using the applied Kaplan-Meier methodology.

17. Secondary Outcome: Part 1b: OS in Participants With TP53 WT Neuroblastoma
Description: as for outcome 16
Time Frame: Up to approximately 29 months
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 2 | 3 | 4
months | NA [NA to NA] — The median and upper and lower limit of the 95% CI was not estimable because there was an insufficient number of events. | 3.2 [1.6 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | NA [1.5 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events.

18. Secondary Outcome: Part 1a: ORR Irrespective of TP53 Status in Participants With Solid Tumor From SE Population According to RECIST v1.1 or INRC
Description: ORR was defined as the percentage of participants with CR or PR at any time during study treatment, on two consecutive occasions >= 4 weeks apart, as determined by the investigator according to RECIST v1.1 or INRC. Per RECIST, CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. Participants who had neuroblastoma were assessed by INRC. Per INRC, CR= <10 mm residual soft tissue at primary site and complete resolution of MIBG or FDG-PET uptake at primary site. PR= ≥ 30% decrease in longest diameter of primary site and MIBG or FDG-PET uptake at primary site stable, improved, or resolved. Soft tissue & bone metastases: CR= resolution of all disease sites; PR= ≥30% decrease in sum of non-primary target lesions, with no new lesions or ≥50% reduction in MIBG score or in number of FDG-PET-avid bone lesions; Bone marrow: CR= no tumor infiltration on reassessment.
Time Frame: From screening (maximum 28 days) up to Cycle 5 (cycle length=28 days)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg
Number analyzed (Participants) | 8 | 3 | 6 | 3 | 6
percentage of participants | 0 [0.00 to 36.94] | 0 [0.00 to 70.76] | 0 [0.00 to 45.93] | 0 [0.00 to 70.76] | 0 [0.00 to 45.93]

19. Secondary Outcome: Part 1b: ORR Irrespective of TP53 Status in Participants With Neuroblastoma From SE Population According to INRC
Description: ORR was defined as the percentage of participants with CR or PR at any time during study treatment, on 2 consecutive occasions ≥ 4 weeks apart, as determined by the investigator per INRC. Primary tumor: CR= <10 mm residual soft tissue at primary site and complete resolution of MIBG or FDG-PET uptake at primary site. PR= ≥ 30% decrease in longest diameter of primary site and MIBG or FDG-PET uptake at primary site stable, improved, or resolved. Soft tissue & bone metastases: CR= resolution of all disease sites; PR= ≥30% decrease in sum of non-primary target lesions, with no new lesions or ≥50% reduction in MIBG score or in number of FDG-PET-avid bone lesions; Bone marrow: CR= no tumor infiltration on reassessment. Percentages have been rounded off to nearest decimal point.
Time Frame: From screening (maximum 28 days) up to Cycle 6 (cycle length=28 days)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 0 [0.00 to 70.76] | 33.3 [0.84 to 90.57] | 0 [0.00 to 45.93]

20. Secondary Outcome: Part 1a: Maximum Plasma Concentration (Cmax) of Idasanutlin as a Monotherapy
Time Frame: Days 1 and 5 of Cycle 1 (cycle length = 28 days)
Population: Pharmacokinetic (PK)-evaluable population included all participants who received at least one dose of study treatment and who have data from at least one post dose sample. One participant assigned to the 6.4 mg/kg dose level received a dose of 3.8 mg/kg due to the maximum absolute dose cap of 300 mg/day in protocol v3 and earlier. Hence this participant has been reported in a separate arm for PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL(nanograms/millilitres)
Groups:
- Part 1a: Idasanutlin 3.8 mg/kg: Participants with solid tumors received idasanutlin 3.8 mg/kg orally QD on Days 1-5 of each 28-day cycle until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 3.8 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg
Number analyzed (Participants) | 8 | 3 | 1 | 6 | 2 | 6
ng/mL(nanograms/millilitres)
  Cycle 1 Day 1 | 1429 (36) | 2110 (27) | 1560 (NA) — Since only 1 participant was analyzed Geometric Coefficient of Variation was not estimable. | 3174 (25) | 4474 (90) | 5102 (67)
  Cycle 1 Day 5 | 2548 (21) | 2784 (27) | 2940 (NA) — Since only 1 participant was analyzed Geometric Coefficient of Variation was not estimable. | 4892 (53) | 7748 (81) | 6298 (67)

21. Secondary Outcome: Part 1b: Cmax of Idasanutlin in Combination With Chemotherapy or Venetoclax
Time Frame: Days 1 and 5 of Cycle 1 (cycle length = 28 days)
Population: PK-evaluable population included all participants who received at least one dose of study treatment and who have data from at least one post dose sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy: Participants with neuroblastoma received idasanutlin 3.6 mg/kg orally in combination with cyclophosphamide 250 mg/m^2 and topotecan 0.75 mg/m^2 as an IV infusion QD on Days 1-5 of each 28-day cycle. Treatment was administered until disease progression, death, unacceptable toxicity, or decision to discontinue, whichever occurred first.
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 3 | 3 | 6
ng/mL
  Cycle 1 Day 1 | 2834 (31) | 1540 (11) | 2131 (43)
  Cycle 1 Day 5 | 2393 (32) | 2110 (72) | 2272 (32)

22. Secondary Outcome: Part 1a: Cmax of Idasanutilin Metabolite M4 Following Idasanutilin as a Monotherapy
Time Frame: Days 1 and 5 of Cycle 1 (cycle length = 28 days)
Population: PK-evaluable population included all participants who received at least one dose of study treatment and who have data from at least one post dose sample. One participant assigned to the 6.4 mg/kg dose level received a dose of 3.8 mg/kg due to the maximum absolute dose cap of 300 mg/day in protocol v3 and earlier. Hence this participant has been reported in a separate arm for PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 3.8 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg
Number analyzed (Participants) | 8 | 3 | 1 | 6 | 2 | 6
ng/mL
  Cycle 1 Day 1 | 129 (63) | 184 (39) | 72 (NA) — Since only 1 participant was analyzed Geometric Coefficient of Variation was not estimable. | 340 (60) | 542 (153) | 575 (148)
  Cycle 1 Day 5 | 436 (73) | 419 (23) | 345 (NA) — Since only 1 participant was analyzed Geometric Coefficient of Variation was not estimable. | 820 (76) | 1865 (197) | 1511 (201)

23. Secondary Outcome: Part 1b: Cmax of Idasanutlin Metabolite M4 (Idasanutilin in Combination With Chemotherapy or Venetoclax)
Time Frame: Days 1 and 5 of Cycle 1 (cycle length = 28 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 3 | 3 | 6
ng/mL
  Cycle 1 Day 1 | 229 (56) | 214 (72) | 213 (67)
  Cycle 1 Day 5 | 442 (148) | 524 (97) | 369 (58)

24. Secondary Outcome: Part 1b: Plasma Concentration of Venetoclax in Combination With Idasanutlin
Time Frame: Cycle 1: Predose on Days 2 and 5, 4 and 6 hours post dose on Days 1 and 5 (1 cycle = 28 days)
Population: PK-evaluable population included all participants who received at least one dose of study treatment and who have data from at least one post dose sample. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
Number analyzed (Participants) | 6
ng/mL
  Cycle 1 Day 1, Post dose 4 Hours | 693 (44)
  Cycle 1 Day 1, Post dose 6 Hours: number analyzed (Participants) | 5
  Cycle 1 Day 1, Post dose 6 Hours | 669 (86)
  Cycle 1 Day 2, Predose | 202 (109)
  Cycle 1 Day 5, Predose | 221 (108)
  Cycle 1 Day 5, Post dose 4 Hours | 1145 (45)
  Cycle 1 Day 5, Post dose 6 Hours | 968 (39)

25. Secondary Outcome: Parts 1, 2 and 3: Number of Participants With Leukemia Receiving Transplant After Study Treatment
Time Frame: Up to approximately 29 months
Population: The study was terminated before initiation of Parts 2 and 3 as per sponsor's decision. No participants with leukemia were enrolled in Part 1. Hence no data were collected, and this outcome measure was not assessed or analyzed.
Groups:
- Part 1 (Leukemia): Participants with AML and ALL were planned to be enrolled in various cohorts in Part 1. Participants with AML and ALL were to receive idasanutlin in combination venetoclax 400 mg. Participants with AML were to receive idasanutlin plus fludarabine 30 mg/m^2 and high dose cytarabine 2000 mg/m^2 (FLA) on Days 1-5 of each 28-day cycle.
- Part 2 (Leukemia): Participants with AML or ALL were planned to be enrolled in various cohorts in Part 2. Participants with AML were to receive idasanutlin plus fludarabine 30 mg/m^2 and high dose cytarabine 2000 mg/m^2 (FLA) on Days 1-5 of each 28-day cycle. Participants with ALL were to receive idasanutlin plus venetoclax 600 mg on Days 1-5 of each 28-day cycle.
- Part 3: Expansion (Leukemia): Potential expansion of idasanutlin combination cohorts for participants with TP35 WT AML or ALL from Part 1b and 2 meeting the pre-defined efficacy criteria were planned to be initiated in Part 3.
Arm/Group | Part 1 (Leukemia) | Part 2 (Leukemia) | Part 3: Expansion (Leukemia)
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Parts 1, 2 and 3: Duration of Objective Response in Participants With Leukemia
Description: DOR, defined as the time from the first tumor assessment that supports the participant's objective response (CR, CRp, CRi) to the time of relapse, or death from any cause, whichever occurs first. CR=Bone marrow blasts <5% (AML) and no evidence of circulating blasts, must be <1% (ALL); absence of blasts with Auer rods (AML); absence of extramedullary disease; absolute neutrophil count (ANC) >1.0*10^9/L [1000µL]; platelet count > 100*10^9/L (100,000/µL); independence of transfusions for a minimum of 1 week (AML and ALL). CRi= All CR criteria except for ANC <1.0*10^9/L[1000/µL] or insufficient recovery of platelet count <100* 10^9/L [100,000/µL] (AML and ALL). CRp=All CR criteria except for ANC >1.0*10^9/L[1000/µL]) or but with insufficient recovery of platelet (<100* 10^9/L [100,000/µL]) (ALL). Relapse=participants who achieved a CR/CRp/CRi & subsequently developed: Bone marrow blasts ≥5%; reappearance of blasts in the blood ≥1%; or development of extra-medullary disease.
Time Frame: Up to approximately 29 months
Population: as for outcome 25
Groups:
- Part 1 (Leukemia): Participants with AML or ALL were planned to be enrolled in various cohorts in Part 1. Participants with AML or ALL were to receive idasanutlin in combination venetoclax 400 mg. Participants with AML were to receive idasanutlin plus fludarabine 30 mg/m^2 and high dose cytarabine 2000 mg/m^2 (FLA) on Days 1-5 of each 28-day cycle.
Arm/Group | Part 1 (Leukemia) | Part 2 (Leukemia) | Part 3: Expansion (Leukemia)
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Parts 1, 2 and 3: Event-Free Survival (EFS) in Participants With Leukemia
Description: EFS=time from initiation of study drug to first documented occurrence of M3 marrow after Cycle 1, failure to achieve CR/CRp/CRi after Cycle 2, disease progression, relapse after achieving CR/CRp/CRi, or death from any cause, whichever occurs first. CR=Bone marrow blasts <5% (AML) & no evidence of circulating blasts, must be <1% (ALL); absence of blasts with Auer rods (AML); absence of extramedullary disease; ANC >1.0*10^9/L [1000µL]; platelet count > 100*10^9/L (100,000/µL); no transfusions for a minimum of 1 week (AML & ALL). CRi= All CR criteria except for ANC <1.0*10^9/L[1000/µL] or insufficient recovery of platelet count <100* 10^9/L [100,000/µL] (AML & ALL). CRp=All CR criteria except for ANC >1.0*10^9/L[1000/µL]) or but with insufficient recovery of platelet (<100* 10^9/L [100,000/µL]) (ALL). Relapse=participants who achieved a CR/CRp/CRi & subsequently developed: Bone marrow blasts ≥5%; reappearance of blasts in blood ≥1%; or development of extra-medullary disease.
Time Frame: Up to approximately 29 months
Population: as for outcome 25
Arm/Group | Part 1 (Leukemia) | Part 2 (Leukemia) | Part 3: Expansion (Leukemia)
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Parts 1, 2 and 3: OS in Participants With Leukemia
Description: OS was defined as the time from initiation of study drug to death from any cause.
Time Frame: Up to approximately 29 months
Population: The study was terminated before initiation of Part 2 and 3 as per sponsor's decision. No participants with leukemia were enrolled in Part 1. Hence no data were collected, and this outcome measure was not assessed or analyzed.
Arm/Group | Part 1 (Leukemia) | Part 2 (Leukemia) | Part 3: Expansion (Leukemia)
Number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: Parts 1, 2 and 3: CRR of Efficacy-evaluable Population Irrespective of TP53 Status in Participants With Leukemia
Description: CRR was defined as the percentage of participants with CR, CRi, or CRp within 2 cycles of study treatment. CR=Bone marrow blasts <5% (AML) and no evidence of circulating blasts, must be <1% (ALL); absence of blasts with Auer rods (AML); absence of extramedullary disease; absolute neutrophil count (ANC) >1.0*10^9/L [1000/µL]; platelet count > 100*10^9/L (100,000/µL); independence of transfusions for a minimum of 1 week (AML and ALL). CRi= All CR criteria except for ANC <1.0*10^9/L[1000/µL] or insufficient recovery of platelet count <100* 10^9/L [100,000/µL] (AML and ALL). CRp=All CR criteria except for ANC >1.0*10^9/L[1000/µL]) or but with insufficient recovery of platelet (<100* 10^9/L [100,000/µL]) (ALL).
Time Frame: Up to approximately 29 months
Population: as for outcome 28
Arm/Group | Part 1 (Leukemia) | Part 2 (Leukemia) | Part 3: Expansion (Leukemia)
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Parts 1, 2 and 3: MRD - Negative Rate in Participants With ALL
Description: MRD - negative rate was defined as defined as the percentage of participants with AML who are MRD negative within 2 cycles of study treatment.
Time Frame: Up to approximately 29 months
Population: as for outcome 25
Groups:
- Part 1 (ALL): Participants with ALL were planned to be enrolled in various cohorts in Part 1 and receive idasanutlin in combination venetoclax 400 mg.
- Part 2 (ALL): Participants with ALL were planned to be enrolled in Part 2 and receive idasanutlin plus venetoclax 600 mg on Days 1-5 of each 28-day cycle.
- Part 3: Expansion (ALL): Potential expansion of idasanutlin combination cohorts for participants with TP35 WT ALL from Part 1b and 2 meeting the pre-defined efficacy criteria were planned to be initiated in Part 3.
Arm/Group | Part 1 (ALL) | Part 2 (ALL) | Part 3: Expansion (ALL)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: From screening up to 30 days after study treatment discontinuation (approximately 7 months) All-cause mortality: From screening up to end of follow up (approximately 29 months)
Description: Safety population. One participant enrolled in idasanutlin 6.4 mg/kg cohort received a dose of 3.8 mg/kg due to maximum dose capping of 300 mg/day in protocol v3. As pre-planned, for safety evaluation and as part of the modified continual reassessment method of escalation with overdose control (mCRM) review, this participant was considered to be a part of the 6.4 mg/kg cohort in which the participant was enrolled. Thus, AEs for this participant are included in the 6.4 mg/kg cohort.
Arm/Group | Part 1a: Idasanutlin 2 mg/kg | Part 1a: Idasanutlin 3 mg/kg | Part 1a: Idasanutlin 4.5 mg/kg | Part 1a: Idasanutlin 6.4 mg/kg | Part 1a: Idasanutlin 8 mg/kg | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6 mg/kg) +Chemotherapy | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax
All-Cause Mortality (participants affected / at risk) | 8/8 | 3/3 | 6/6 | 2/3 | 5/6 | 0/3 | 2/3 | 3/6
Serious Adverse Events (participants affected / at risk) | 6/8 | 3/3 | 4/6 | 2/3 | 6/6 | 2/3 | 3/3 | 4/6
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 6/6 | 3/3 | 6/6 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a: Idasanutlin 2 mg/kg (N=8) | Part 1a: Idasanutlin 3 mg/kg (N=3) | Part 1a: Idasanutlin 4.5 mg/kg (N=6) | Part 1a: Idasanutlin 6.4 mg/kg (N=3) | Part 1a: Idasanutlin 8 mg/kg (N=6) | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy (N=3) | Part 1b: Idasanutlin (3.6 mg/kg) +Chemotherapy (N=3) | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (6) | 2 (3) | 2 (3) | 1 (1) | 3 (5) | 1 (1) | 2 (3) | 0 (0)
Hematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (7) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a: Idasanutlin 2 mg/kg (N=8) | Part 1a: Idasanutlin 3 mg/kg (N=3) | Part 1a: Idasanutlin 4.5 mg/kg (N=6) | Part 1a: Idasanutlin 6.4 mg/kg (N=3) | Part 1a: Idasanutlin 8 mg/kg (N=6) | Part 1b: Idasanutlin (2.8mg/kg) +Chemotherapy (N=3) | Part 1b: Idasanutlin (3.6 mg/kg) +Chemotherapy (N=3) | Part 1b: Idasanutlin (3.6mg/kg) + Venetoclax (N=6)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 3 (4) | 1 (1) | 6 (6) | 3 (4) | 3 (9) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (3) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (10) | 2 (3) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 3 (7) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (3) | 5 (7) | 3 (4) | 1 (1) | 1 (1) | 2 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (6) | 4 (6) | 2 (2) | 3 (3) | 0 (0) | 2 (5) | 5 (6)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (7) | 2 (8) | 4 (9) | 1 (3) | 2 (2) | 1 (1) | 2 (7) | 4 (7)
Asthenia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (5) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (6) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (9) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (5) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04029688/Prot_SAP_000.pdf